CLINICAL TRIAL: NCT02525068
Title: A Randomised Phase II Study of Enzalutamide (MDV3100) in Combination With AZD5363 in Patients With Metastatic Castration-Resistant Prostate Cancer (RE-AKT)
Brief Title: A Study of Enzalutamide in Combination With AZD5363 in Patients With mCRPC
Acronym: RE-AKT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICR-CTSU/2012/10037; 2013-004091-34 (EudraCT Number); CRUKE/12/050 (Other Grant/Funding Number: Cancer Research UK); ISRCTN17168679 (Registry Identifier: Randomised Controlled Trials); ISS53630011 (Other Grant/Funding Number: AstraZenca)
Record Dates: First submitted 2015-07-17; First posted 2015-08-17 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2015-08

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: enzalutamide; AZD5363; Prostate
MeSH Terms: interventions — capivasertib; enzalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase ISafety Run-In (Experimental): 18 patients will receive the combination of enzalutamide and AZD5363 (on an intermittent schedule 4 days on 3 days off) to determine the AZD5363 dose to be used for the randomised phase II and single stage phase II expansion cohort. Approximately three dose-levels of AZD5363 in combination with enzalutamide are planned although other dose levels may be required.
  Interventions: Drug: AZD5363; Drug: Enzalutamide
- Randomised phase II (Placebo Comparator): 100 patients will be randomised in a 1:1 ratio to receive 160mg enzalutamide od + AZD5363 bid 4 days on 3 days off (recommended dose from Phase I) vs 160mg enzalutamide od + matching placebo bid 4 days on 3 days off.
  Interventions: Drug: AZD5363; Drug: Enzalutamide
- Single stage phase II expansion cohort (Experimental): Following progression on enzalutamide alone, 18 patients will receive enzalutamide 160mg od and AZD5363 bid (recommended dose from phase I) 4 days on 3 days off
  Interventions: Drug: AZD5363; Drug: Enzalutamide

INTERVENTIONS:
Drug: AZD5363 — Until confirmed disease progression.
Drug: Enzalutamide — Until confirmed disease progression.
  Other Names: MDV3100; Xtandi

SUMMARY:
A multicentre prospective, randomised, phase II interventional study in mCRPC patients previously treated with 1-2 lines of chemotherapy and at least 12 weeks of abiraterone with a safety run-in and single stage phase II expansion cohort.

DETAILED DESCRIPTION:
Patients with mCRPC will receive enzalutamide and AZD5363 (or enzalutamide and placebo in the randomised phase II) until confirmed disease progression.

The trial aims to identify the safety and tolerability of enzalutamide and AZD5363 and identify recommended phase II dose of AZD5363 (phase I safety run-in). The randomised phase II will estimate and compare the anti-tumour activity of AZD5363 and enzalutamide, and placebo and enzalutamide as measured by response. The single stage phase II expansion cohort will estimate the anti-tumour activity of AZD5363 and enzalutamide in patients who have previously progressed on enzalutamide alone.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Histological diagnosis of adenocarcinoma of the prostate and with tumour tissue accessible for research analyses for this trial (e.g. Phosphatase and Tensin Homologue (PTEN) testing). Patients who have no histological diagnosis must be willing to undergo a biopsy to prove prostate adenocarcinoma.
3. Metastatic Castration-Resistant Prostate Cancer (mCRPC).
4. Progressed after 1 or 2 lines of taxane based chemotherapy.
5. Progressed after abiraterone (pre or post chemotherapy). Patients must have received at least 12 weeks of treatment with abiraterone.
6. Age ≥18 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
8. PSA ≥ 10ng/ml.
9. Documented willingness to use an effective means of contraception while participating in the study and for 12 months post last dose of treatment
10. Documented ongoing castrate serum testosterone <50 ng/dL (<2.0 nM).
11. Received prior castration by orchiectomy and/or ongoing Luteinizing Hormone-Releasing Hormone (LH-RH) agonist treatment.
12. Progression of disease by PSA utilizing PCWG2 criteria and at least another of the following criteria;

    1. Bone scan: disease progression as defined by at least 2 new lesions on bone scan.
    2. Soft tissue disease progression defined by modified RECIST 1.1.
    3. Clinical progression with worsening pain and the need for palliative radiotherapy for bone metastases.

    PHASE I SAFETY RUN IN and EXPANSION COHORT - inclusion criteria:
13. Willing to have a biopsy to obtain tumour tissue for biomarker analyses prior to and after treatment.

    SINGLE STAGE PHASE II EXPANSION COHORT ONLY - inclusion criteria:
14. Prior exposure to enzalutamide of at least 12 weeks is required with documented disease progression biochemically and/or radiologically by PCWG2 or RECIST 1.1 criteria. Patients should have received at least 12 weeks of enzalutamide outside of the trial with evidence of disease progression (by PSA with 3 rising values as per PCWG2 criteria or soft tissue progression as per RECIST v1.1).
15. Archival tumour tissue available for the analysis of PTEN loss by the central laboratory

Exclusion Criteria:

1. Prior treatment with enzalutamide (MDV3100) (not applicable for the phase I safety run in or for the single stage phase II expansion cohort, see inclusion criteria 14).
2. Prior treatment with Phosphatidylinositide 3-kinases (PI3K), AKT, TOR kinase or Mammalian target of rapamycin (mTOR) inhibitors (see Appendix C).
3. Surgery, chemotherapy, or other anti-cancer therapy within 4 weeks prior to trial entry/randomisation into the study (6 weeks for bicalutamide). Any other therapies for prostate cancer, other than Gonadotropin-releasing hormone (GnRH) analogue therapy, such as progesterone, medroxyprogesterone, progestins (megestrol), or 5-alpha reductase inhibitors (e.g., finasteride or dutasteride), must be discontinued at least 2 weeks before the first dose of study drug.
4. Participation in another clinical trial and any concurrent treatment with any investigational drug within 4 weeks prior to trial entry / randomisation.
5. Prior limited field radiotherapy within 2 weeks or wide field radiotherapy within 4 weeks of trial entry / randomisation.
6. History of seizure or any condition that may predispose to seizure including, but not limited to underlying brain injury, stroke, primary brain tumours, brain metastases, or alcoholism.
7. History of loss of consciousness or transient ischemic attack within the previous 12 months of trial entry / randomisation.
8. Known brain or leptomeningeal involvement.
9. Use of potent inhibitors or inducers of Cytochrome P450 isoenzymes (CYP3A4, CYP2C9, CYP2C19 and CYP2D6) (see Appendix B) within 2 weeks before trial entry / randomisation (3 weeks for St John's Wort) must be avoided.
10. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

    1. Diagnosis of diabetes mellitus type I
    2. Fasting plasma glucose ≥ 7.0 mmol/L for those patients without a pre-existing diagnosis of Type 2 diabetes mellitus

       ≥ 9.3 mmol/L for those patients with a pre-existing diagnosis of Type 2 diabetes mellitus
    3. Glycosylated haemoglobin (HbA1C) ≥8.0% at screening (63.9 mmol/mol) (conversion equation for HbA1C [IFCC-HbA1C (mmol/mol) = [DCCT-HbA1C (%) - 2.15] x 10.929)
    4. Requirement for insulin for routine diabetic management and control
    5. Requirement for more than two oral hypoglycaemic medications for routine diabetic management and control
11. Inadequate organ and bone marrow function as evidenced by:

    1. Haemoglobin <85 g/L
    2. Absolute neutrophil count <1.0 x 109/L
    3. Platelet count < 75 x 109/L
    4. Albumin ≤25 g/dL
    5. Aspartate Transaminase (AST) / Serum Glutamic-Oxaloacetic Transaminase (SGOT) and/or Alanine Transaminase (ALT) / Serum Glutamic Pyruvate Transaminase (SGPT) ≥ 2.5 x Upper Limit of Normal (ULN) (≥ 5 x ULN if liver metastases present)
    6. Total bilirubin ≥ 1.5 x ULN (except for patient with documented Gilbert's disease)
    7. Serum Creatinine > 1.5 x ULN
12. Inability or unwillingness to swallow oral medication.
13. Malabsorption syndrome or other condition that would interfere with enteral absorption.
14. Any of the following cardiac criteria;

    1. Mean resting corrected QT interval (QTcF) >470msec obtained from 3 consecutive ECGs taken within 5 minutes
    2. Any clinically important abnormalities in rhythm, conduction, or morphology of a resting ECG (e.g., complete left bundle branch block, third degree heart block)
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval or with a potential for Torsades de Pointes
    4. Experience of any of the following procedures or conditions in the preceding six months:coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association (NYHA) ≥ Grade2
    5. Uncontrolled hypotension defined as - systolic blood pressure (BP) <90 mmHg and/or diastolic BP <50 mmHg
15. Clinically significant history of liver disease consistent with Child-Pugh Class B or C, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
16. Any other finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patients at high risk from treatment complications.
17. Need for chronic corticosteroid therapy of >10 mg of prednisolone or >0.5mg of dexamethasone per day or an equivalent dose of other anti-inflammatory corticosteroid, for the use of concomitant steroids on this trial please refer to section 12.1. Patients in which corticosteroids cannot be stopped prior to entering the trial are allowed a maximum of 10mg of prednisolone per day or equivalent. In the case of corticosteroid discontinuation, a 2-week (14 days) washout is required with a mandatory PSA check prior to starting the trial. If the PSA has declined compared to the value obtained prior to stopping corticosteroids, patients will not be eligible for study. Patients can only enter the study with a confirmed PSA increase.
18. Malignancies other than prostate cancer within 5 years prior to trial entry / randomisation, except for adequately treated basal or squamous cell skin cancer.
19. Unresolved clinically significant toxicity from prior therapy except for alopecia and Grade 1 peripheral neuropathy.
20. Inability to comply with study and follow-up procedures.
21. Patients with predominately small cell or neuroendocrine differentiated prostate cancer are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Phase I: Type, frequency, severity, seriousness and relatedness of adverse events | 35 days
  Type according to Medical Dictionary for Regulatory Activities (MedDRA), frequency according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4, seriousness, and relatedness of study treatment-emergent adverse events will be assessed
Phase I: Laboratory abnormalities will be assessed according to NCI CTCAE v4 | 35 days
Randomised phase II: Best overall tumour response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to an estimated 22-24 months
  Best overall tumour response as defined by Prostate Specific Antigen (PSA) decline of ≥50% (according to PCWG2), confirmed objective response by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 or ONLY for patients with detectable circulating tumour cell count of ≥5/7.5ml blood at baseline, conversion of CTC <5/7.5ml blood nadir
Phase II expansion: Best overall tumour response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to an estimated 22-24 months
  Best overall tumour response as defined by PSA decline of ≥50% (according to PCWG2), confirmed objective response by RECIST 1.1 or ONLY for patients with detectable circulating tumour cell count of ≥5/7.5ml blood at baseline, conversion of CTC <5/7.5ml blood nadir

SECONDARY OUTCOMES:
Phase I and phase II expansion only - Pharmacokinetic (PK) assay analyses | 35 days
  PK assay analysis including endpoints of Peak Plasma Concentration (Cmax) and Area under the plasma concentration versus time curve (AUC)
Phase I - Antitumour activity of the combination | 35 days
Randomised phase II and phase II expansion - Overall survival and radiographic progression free survival | From date of randomization/trial entry until the date of first documented progression or date of death from any cause, whichever came first, assessed up to (estimated) 12 months
Maximum PSA decline and circulating tumour cell (CTC) fall | 12 weeks
  Maximum PSA decline and CTC fall by 30% at any time during the trial and at 12 weeks.
Pain Palliation - Randomised phase II only | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to (estimated) 12 months
  Pain palliation will be assessed using the Brief Pain Inventory (Short Form) (BPI-SF) worst pain intensity score
Number of Adverse events will be graded according to NCI-CTCAE v4 | From trial entry until 30 days post date of last dose or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Johann De Bono, Professor, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Kolinsky MP, Rescigno P, Bianchini D, Zafeiriou Z, Mehra N, Mateo J, Michalarea V, Riisnaes R, Crespo M, Figueiredo I, Miranda S, Nava Rodrigues D, Flohr P, Tunariu N, Banerji U, Ruddle R, Sharp A, Welti J, Lambros M, Carreira S, Raynaud FI, Swales KE, Plymate S, Luo J, Tovey H, Porta N, Slade R, Leonard L, Hall E, de Bono JS. A phase I dose-escalation study of enzalutamide in combination with the AKT inhibitor AZD5363 (capivasertib) in patients with metastatic castration-resistant prostate cancer. Ann Oncol. 2020 May;31(5):619-625. doi: 10.1016/j.annonc.2020.01.074. Epub 2020 Feb 21. PMID 32205016